CLINICAL TRIAL: NCT02950506
Title: Transcranial Direct Current Stimulation and Cognitive Remediation Therapy for Interictal Dysfunction in Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CTSI24219
Record Dates: First submitted 2016-08-10; First posted 2016-11-01 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Epilepsy
Keywords: Interictal; Cognitive; Dysfunction; tDCS; transcranial direct current stimulation
MeSH Terms: conditions — Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Active Comparator): There will be a total of 14 visits in the study: will complete a screening visit, an initial visit, 10 session visits with active tDCS(transcranial direct current stimulation) andcognitive remediation therapy, and follow--up visits immediately (within 5 days), 1 and 3 months after the last intervention. Subjects will be informed of their group assignment at the end of the study.
  Interventions: Device: transcranial direct current stimulation; Other: Cognitive Remediation Therapy
- Sham tDCS (Sham Comparator): There will be a total of 14 visits in the study: will complete a screening visit, an initial visit, 10 session visits with sham tDCS and cognitive remediation therapy, and follow--up visits immediately (within 5 days), 1 and 3 months after the last intervention. Subjects will be informed of their group assignment at the end of the study.
  Interventions: Other: Cognitive Remediation Therapy

INTERVENTIONS:
Device: transcranial direct current stimulation — The anode will be placed over left DLPFC at F3, according to the 10-20 international system for EEG electrode placement. The cathode will be placed over the contralateral supraorbital area. They will be placed via two saline soaked electrode sponges (3 cm x 4.5 cm).After electrodes have been placed, the participants will be instructed to log into CRT software using a unique patient identifier. The CRT software that will be used will be Cogmed working memory training program (Pearson Education, Inc.)Active tDCS will be applied at a ramp-like fashion from 0 to 2mA over 10 seconds, and will be ramped down for the last 10 seconds of stimulation. Active tDCS will last 20 minutes each session. The sham procedure involves only 30 seconds of stimulation at 2mA.
  Other Names: tDCS; Starstim; Starstim Enobio; Starstim 20; Starstim Enobio 20; Neuroelectrics Starstim
  Arms: Active tDCS
Other: Cognitive Remediation Therapy — The CRT software that will be used will be Cogmed working memory training program (Pearson Education, Inc.). Cogmed is a targeted computerized training program that has been shown to improve working memory and attention. (Spencer-Smith 2015).
  Other Names: CRT; Cogmed

SUMMARY:
The purpose of this study is to investigate whether tDCS enhances the effect of cognitive remediation therapy on cognition and functional outcome in patients with epilepsy. There has been evidence that working memory performance is enhanced in healthy subjects. Acute tDCS studies have found improvements in working memory performance in subjects with other neurological diseases. To date, there have been no published studies examining whether can enhance learning during multi-session cognitive remediation over 2 weeks in subjects with epilepsy. This study could have potential application as a non-invasive clinical intervention for interictal dysfunction in epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurological disorder affecting 50 million people worldwide. Patients suffer not only from recurring seizures, but also from cognitive deficits despite adequate treatment control. Cognitive remediation therapy (CRT) is a therapeutic intervention that has recently shown promise in improving cognitive impairment in many neuropsychological disorders. Transcranial direct current stimulation (tDCS) is a non-invasive method that modulates cortical excitability. It works by applying weak electrical currents to the scalp that induce acute modifications of neuronal membrane potentials, producing long-lasting changes in the bioelectric activity of underlying brain tissue. It is postulated that tDCS enhances benefit gained through cognitive remediation therapy. These interventions have yet to be combined with each other for the treatment of interictal dysfunction in patients with epilepsy. The goal of the study is to investigate whether the introduction of tDCS in addition to CRT is effective in the treatment of cognitive impairment in patients suffering from epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Epilepsy diagnosis confirmed by the UMN Comprehensive Epilepsy Center
* Complete seizure logs of the type in standard clinic use at the UMN Comprehensive Epilepsy Center for at least 12 weeks prior to study entry
* Stable CNS medications for the 2 weeks prior to the initiation visit and expected to continue with current medication doses for the two weeks of the intervention
* No diagnosis of mental retardation (IQ not less than 70) or pervasive developmental disorder
* At least one subtest of learning and memory less than --1.5 SD
* Sufficient spoken English so as to be able to comprehend testing procedures
* Competent and willing to provide consent

Exclusion Criteria:

* Occurrence of generalized convulsive status epilepticus or of complex partial status epilepticus within 1 year prior to study entry
* Occurrence of more than 1 generalized tonic-clonic (GTC) seizure per month, or more than 4 complex partial (CP) seizures per week, as reported in the subject's seizure logs for 12 weeks prior to study entry
* Occurrence of GTC seizure within 48 hours before testing
* Any anti-epileptic medication changes or hospitalizations in the previous 4 weeks
* Additional neurologic disorder other epilepsy and cognitive dysfunctions
* History of metallic cranial plates, screws, or implanted devices
* History of craniotomy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Cogstate Brief Battery | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  The Cogstate Battery is a computerized cognitive assessment program which measures a wide
  range of cognitive functions (e.g. psychomotor speed, reaction time, working memory, divided
  attention, learning), which can be repeated with little to none observed practice effects (Falleti
  2006). All tasks within the battery were adaptations of standard neuro-psychological and
  experimental psychological tests. Time to administer requires approximately 15-20 minutes
  consists of 8 tasks in the form of card games that are presented in succession.
Rey Auditory Verbal Learning Test (AVLT) | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  The Rey Auditory Verbal Learning Test (AVLT) is a measure of immediate auditory and verbal
  memory as well as delayed recall. Participants are given a list of 15 unrelated words repeated
  over five different trials and are asked to repeat. Another list of 15 unrelated words are given and
  the client must again repeat the original list of 15 words and then again after 30 minutes.
  Approximately 45-50 minutes is required for the procedure. (Loring et al. 2008, Strauss 2006)
Picture Sequence Memory Test | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  The Picture Sequence Memory Test (PSMT) is a measure for use in the assessment of episodic
  memory. Participants are asked to recall, in increasing length, a series of illustrated objects and
  activities that are presented in a particular order on the computer screen. The participants are
  asked to recall the sequence of pictures that is demonstrated over two learning trials. The number
  of pictures may vary depending on the age. The test takes approximately 7 minutes to administer.
  (Dikmen et al. 2014)
Flanker Inhibitory Control and Attention Task | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  This task measures both a participant's attention and inhibitory control. The test requires the
  participant to focus on a given arrow while inhibiting attention to other arrows surrounding it.
  (Heaton et al. 2014) Sometimes the middle stimulus is pointing in the same direction as the
  "flankers" (congruent) and sometimes in the opposite direction (incongruent). Scoring is based
  on a combination of accuracy and reaction time. The test takes approximately 3 minutes to
  administer.
Dimensional Change Card Sort Test | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  DCCS is an assessment to measure of cognitive flexibility. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension(e.g., shape). "Switch" trials are also employed, in which the participant must change the dimension being matched. For example, after 4 straight trials matching on shape,the participant may be asked to match on color on the next trial and then go back to shape, thus requiring the cognitive flexibility to quickly choose the correct stimulus. Scoring is based on a combination of accuracy and reaction time. This test takes approximately 4 minutes to administer.

SECONDARY OUTCOMES:
Oral Symbol Digit Test | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  This instrument is a measure of processing speed. (Denboer et al. 2014). The participant is presented with a set of nine symbols on the computer screen, each associated with a number 1-9, and is then presented with a series of symbols without numbers and is asked to orally say each number that should go with that symbol, without skipping any. The score is equal to the number of symbols correctly identified orally within two minutes. This takes approximately 3 minutes.
Cogstate Brief Battery | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  The Cogstate Battery is a computerized cognitive assessment program which measures a wide
  range of cognitive functions (e.g. psychomotor speed, reaction time, working memory, divided
  attention, learning), which can be repeated with little to none observed practice effects (Falleti
  2006). All tasks within the battery were adaptations of standard neuro-psychological and
  experimental psychological tests. Time to administer requires approximately 15-20 minutes
  consists of 8 tasks in the form of card games that are presented in succession.
Quality of Life | Change from baseline to 5 days, 1 month, and 3 months after last intervention visit.
  To asses quality of life the Quality of Life in Epilepsy Inventory 31 will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Henry, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Comprehensive Epilepsy Center(MINCEP), Saint Louis Park, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available.

REFERENCES:
- [Background] Andrews SC, Hoy KE, Enticott PG, Daskalakis ZJ, Fitzgerald PB. Improving working memory: the effect of combining cognitive activity and anodal transcranial direct current stimulation to the left dorsolateral prefrontal cortex. Brain Stimul. 2011 Apr;4(2):84-9. doi: 10.1016/j.brs.2010.06.004. Epub 2010 Jul 11. PMID 21511208
- [Background] Benedict, Ralph H B, David Schretlen, Lowell Groninger, and Jason Brandt. 1998. "Hopkins Verbal Learning Test - Revised: Normative Data and Analysis of Inter-Form and Test-Retest Reliability." The Clinical Neuropsychologist 12 (1): 43-55.
- [Background] Benson N, Hulac DM, Kranzler JH. Independent examination of the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV): what does the WAIS-IV measure? Psychol Assess. 2010 Mar;22(1):121-30. doi: 10.1037/a0017767. PMID 20230158
- [Background] Boggio PS, Ferrucci R, Rigonatti SP, Covre P, Nitsche M, Pascual-Leone A, Fregni F. Effects of transcranial direct current stimulation on working memory in patients with Parkinson's disease. J Neurol Sci. 2006 Nov 1;249(1):31-8. doi: 10.1016/j.jns.2006.05.062. Epub 2006 Jul 14. PMID 16843494
- [Background] Brandt, J. & Benedict, R. (2001). Hopkins Verbal Learning Test-Revised: Professional Manual. PAR: Florida
- [Background] Brunelin J, Mondino M, Haesebaert F, Saoud M, Suaud-Chagny MF, Poulet E. Efficacy and safety of bifocal tDCS as an interventional treatment for refractory schizophrenia. Brain Stimul. 2012 Jul;5(3):431-432. doi: 10.1016/j.brs.2011.03.010. Epub 2011 Apr 24. No abstract available. PMID 22037120
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Cramer JA, Perrine K, Devinsky O, Bryant-Comstock L, Meador K, Hermann B. Development and cross-cultural translations of a 31-item quality of life in epilepsy inventory. Epilepsia. 1998 Jan;39(1):81-8. doi: 10.1111/j.1528-1157.1998.tb01278.x. PMID 9578017
- [Background] Del Felice A, Magalini A, Masiero S. Slow-oscillatory Transcranial Direct Current Stimulation Modulates Memory in Temporal Lobe Epilepsy by Altering Sleep Spindle Generators: A Possible Rehabilitation Tool. Brain Stimul. 2015 May-Jun;8(3):567-73. doi: 10.1016/j.brs.2015.01.410. Epub 2015 Jan 30. PMID 25862600
- [Background] Denboer, John W, Christopher Nicholls, Corrine Corte, and Kali Chestnut. 2014. "National Institutes of Health Toolbox Cognition Battery." Archives of Clinical Neuropsychology: The Official Journal of the National Academy of Neuropsychologists, August. doi:10.1093/arclin/acu033.
- [Background] Dikmen SS, Bauer PJ, Weintraub S, Mungas D, Slotkin J, Beaumont JL, Gershon R, Temkin NR, Heaton RK. Measuring episodic memory across the lifespan: NIH Toolbox Picture Sequence Memory Test. J Int Neuropsychol Soc. 2014 Jul;20(6):611-9. doi: 10.1017/S1355617714000460. Epub 2014 Jun 24. PMID 24960230
- [Background] Engelberts NH, Klein M, Ader HJ, Heimans JJ, Trenite DG, van der Ploeg HM. The effectiveness of cognitive rehabilitation for attention deficits in focal seizures: a randomized controlled study. Epilepsia. 2002 Jun;43(6):587-95. doi: 10.1046/j.1528-1157.2002.29401.x. PMID 12060017
- [Background] Falleti MG, Maruff P, Collie A, Darby DG. Practice effects associated with the repeated assessment of cognitive function using the CogState battery at 10-minute, one week and one month test-retest intervals. J Clin Exp Neuropsychol. 2006 Oct;28(7):1095-112. doi: 10.1080/13803390500205718. PMID 16840238
- [Background] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Gazzaley A. Influence of early attentional modulation on working memory. Neuropsychologia. 2011 May;49(6):1410-24. doi: 10.1016/j.neuropsychologia.2010.12.022. Epub 2010 Dec 22. PMID 21184764
- [Background] Haut KM, Lim KO, MacDonald A 3rd. Prefrontal cortical changes following cognitive training in patients with chronic schizophrenia: effects of practice, generalization, and specificity. Neuropsychopharmacology. 2010 Aug;35(9):1850-9. doi: 10.1038/npp.2010.52. Epub 2010 Apr 28. PMID 20428109
- [Background] Heaton RK, Akshoomoff N, Tulsky D, Mungas D, Weintraub S, Dikmen S, Beaumont J, Casaletto KB, Conway K, Slotkin J, Gershon R. Reliability and validity of composite scores from the NIH Toolbox Cognition Battery in adults. J Int Neuropsychol Soc. 2014 Jul;20(6):588-98. doi: 10.1017/S1355617714000241. Epub 2014 Jun 24. PMID 24960398
- [Background] Henry TR, Roman DD. Presurgical epilepsy localization with interictal cerebral dysfunction. Epilepsy Behav. 2011 Feb;20(2):194-208. doi: 10.1016/j.yebeh.2010.12.008. Epub 2011 Jan 22. PMID 21257351
- [Background] Johnson MD, Lim HH, Netoff TI, Connolly AT, Johnson N, Roy A, Holt A, Lim KO, Carey JR, Vitek JL, He B. Neuromodulation for brain disorders: challenges and opportunities. IEEE Trans Biomed Eng. 2013 Mar;60(3):610-24. doi: 10.1109/TBME.2013.2244890. Epub 2013 Feb 1. PMID 23380851
- [Background] Jo JM, Kim YH, Ko MH, Ohn SH, Joen B, Lee KH. Enhancing the working memory of stroke patients using tDCS. Am J Phys Med Rehabil. 2009 May;88(5):404-9. doi: 10.1097/PHM.0b013e3181a0e4cb. PMID 19620953
- [Background] Lin JJ, Mula M, Hermann BP. Uncovering the neurobehavioural comorbidities of epilepsy over the lifespan. Lancet. 2012 Sep 29;380(9848):1180-92. doi: 10.1016/S0140-6736(12)61455-X. PMID 23021287
- [Background] Loring DW, Strauss E, Hermann BP, Barr WB, Perrine K, Trenerry MR, Chelune G, Westerveld M, Lee GP, Meador KJ, Bowden SC. Differential neuropsychological test sensitivity to left temporal lobe epilepsy. J Int Neuropsychol Soc. 2008 May;14(3):394-400. doi: 10.1017/S1355617708080582. PMID 18419838
- [Background] Mattioli F, Bellomi F, Stampatori C, Capra R, Miniussi C. Neuroenhancement through cognitive training and anodal tDCS in multiple sclerosis. Mult Scler. 2016 Feb;22(2):222-30. doi: 10.1177/1352458515587597. Epub 2015 May 26. PMID 26014600
- [Background] Medalia A, Revheim N, & Herlands T. Cognitive remediation for psychological disorders: therapist guide. Treatments that work. Oxford ; New York: Oxford University Press, 2009.
- [Background] Golden, Charles J. 2002. "Stroop Color and Word Test : A Manual for Clinical and Experimental Uses". Wood Dale, IL.
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nowinski CJ, Victorson D, Cavazos JE, Gershon R, Cella D. Neuro-QOL and the NIH Toolbox: implications for epilepsy. Therapy. 2010 Sep 1;7(5):533-540. doi: 10.2217/thy.10.55. PMID 21552344
- [Background] Oliveira JF, Zanao TA, Valiengo L, Lotufo PA, Bensenor IM, Fregni F, Brunoni AR. Acute working memory improvement after tDCS in antidepressant-free patients with major depressive disorder. Neurosci Lett. 2013 Mar 14;537:60-4. doi: 10.1016/j.neulet.2013.01.023. Epub 2013 Jan 28. PMID 23370288
- [Background] Oyegbile TO, Dow C, Jones J, Bell B, Rutecki P, Sheth R, Seidenberg M, Hermann BP. The nature and course of neuropsychological morbidity in chronic temporal lobe epilepsy. Neurology. 2004 May 25;62(10):1736-42. doi: 10.1212/01.wnl.0000125186.04867.34. PMID 15159470
- [Background] Ponds RW, Hendriks M. Cognitive rehabilitation of memory problems in patients with epilepsy. Seizure. 2006 Jun;15(4):267-73. doi: 10.1016/j.seizure.2006.02.011. Epub 2006 Mar 23. PMID 16563809
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Rzezak P, Moschetta SP, Lima E, Castro CX, Vincentiis S, Coan AC, Guerreiro C, Filho GB, Valente KD. Distinct domains of impulsivity are impaired in juvenile myoclonic epilepsy but not in temporal lobe epilepsy. Epilepsy Behav. 2015 Apr;45:44-8. doi: 10.1016/j.yebeh.2015.02.028. Epub 2015 Mar 25. PMID 25819744
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Spencer-Smith M, Klingberg T. Benefits of a working memory training program for inattention in daily life: a systematic review and meta-analysis. PLoS One. 2015 Mar 20;10(3):e0119522. doi: 10.1371/journal.pone.0119522. eCollection 2015. PMID 25793607
- [Background] Strauss E, Sherman E, Spreen O (2006). Rey Auditory Verbal Learning Test. In Compendium of Neuropsychological Tests (3rd Edition) Oxford University Press.776- 807
- [Background] Tam JW, Schmitter-Edgecombe M. The role of processing speed in the Brief Visuospatial Memory Test - revised. Clin Neuropsychol. 2013;27(6):962-72. doi: 10.1080/13854046.2013.797500. Epub 2013 May 20. PMID 23682755
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Slotkin J, Carlozzi NE, Bauer PJ, Wallner-Allen K, Fox N, Havlik R, Beaumont JL, Mungas D, Manly JJ, Moy C, Conway K, Edwards E, Nowinski CJ, Gershon R. The cognition battery of the NIH toolbox for assessment of neurological and behavioral function: validation in an adult sample. J Int Neuropsychol Soc. 2014 Jul;20(6):567-78. doi: 10.1017/S1355617714000320. Epub 2014 Jun 24. PMID 24959840